CLINICAL TRIAL: NCT02782000
Title: The Model and Effect Assessment of Training General Practitioner for Dementia Early Recognition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Sixth Hospital (Other)
Responsible Party: Principal Investigator, Xiaozhen LV, Assistant Researcher, Peking University Sixth Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: SF2016-4-4116
Record Dates: First submitted 2016-05-18; First posted 2016-05-25 (Estimated); Last update posted 2017-12-27 (Actual); Status verified 2017-12

CONDITIONS: Dementia
Keywords: dementia; early recognition; general practitioner; training
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor

ARMS (2):
- Long-term supervision group (Experimental): Firstly, this group will having lessons about dementia early recognition. Second, this group will receive face-to-face supervision and key messages by Wechat about dementia early recognition once a month in the following 6 months.
  Interventions: Other: lessons,long-term supervision and message
- Short-term supervision group (Active Comparator): Firstly, this group will having lessons about dementia early recognition. Second, this group will receive face-to-face supervision and key messages by Wechat about dementia early recognition once a month in the following 3 months.
  Interventions: Other: lessons,short-term supervision and message

INTERVENTIONS:
Other: lessons,long-term supervision and message
  Arms: Long-term supervision group
Other: lessons,short-term supervision and message
  Arms: Short-term supervision group

SUMMARY:
With the number of aged people increasing and the lifespan lengthen, dementia is becoming a great public challenge in China. Early recognition of dementia is crucial to improve the prognosis of dementia patients and decrease the society disease burden. It is a pity that the early recognition rate of dementia is less than 7% in China. Most of the aged people live in the community and general practitioners (GP) in community provide health service much more frequently than other medical workers. It is suggested that GPs should be the best one to screen dementia in its early period. However, most of GPs have not receive any training about dementia early recognition in China. It is imperative and meaningful to provide training to GPs for improve GPs' knowledge and skills about dementia early recognition. How to train GPs for early recognizing dementia and how about the training effect? Which training model may be better? We did not find consistent conclusion about these questions in China. This study aims to set up an effective and convenient model to training GPs in dementia early recognition. A total of 152 GPs in Beijing will be enrolled and be randomly divided into two groups. One group will firstly have lessons about dementia early recognition and then receive face-to-face supervision and key messages by Wechat about dementia early recognition once a month in the following 6 months. Another group will firstly have lessons about dementia early recognition and then receive face-to-face supervision and key messages by Wechat about dementia early recognition once a month in the following 3 months. The score of knowledge and attitude about dementia early recognition, the accuracy of analyzing dementia cases, the usage of dementia screening scales and the referral rate of dementia will be evaluated at different time point respectively. This study will provide evidence for training GPs effectively in dementia early recognition in the future and will promote dementia early recognition in community.

ELIGIBILITY:
Inclusion Criteria:

* General practitioner on-the-job and providing outpatient service
* Can complete the intervention and questionnaire;
* Providing informed consent voluntarily.

Exclusion Criteria:

* General practitioner who may take a long-term vacation during the study
* Providing less than once outpatient service every week;
* Having no condition to use Wechat;
* Refuse to join in this study.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 162 (Actual)
Dates: Start 2016-08-12 (Actual); Primary Completion 2017-03-22 (Actual); Study Completion 2017-07-18 (Actual)

PRIMARY OUTCOMES:
Difference between the change of the score of knowledge about dementia early recognition from baseline to 7th month in the experimental group and that from baseline to 4th month in the active comparator group. | up to 7 months

SECONDARY OUTCOMES:
Difference between the change of the score of attitude about dementia early recognition from baseline to 7th month in the experimental group and that from baseline to 4th month in the active comparator group. | up to 7 months
Difference between the change of the accurate rate of analyzing dementia case from baseline to 7th month in the experimental group and that from baseline to 4th month in the active comparator group. | up to 7 months
Difference between the number of the elderly screened by each general practitioner per month through the study in the experimental group and that in the active comparator group. | up to 7 months

CONTACTS AND LOCATIONS:
Overall Officials: Xiaozhen LV, PhD, Principal Investigator — Peking University Six Hospital

REFERENCES:
- [Derived] Lv X, Zhao M, Li T, Yuan C, Zhang H, Pu C, Li Z, Zhang N, Yu X, Wang H. Effects of an Enhanced Training on Primary Care Providers Knowledge, Attitudes, Service and Skills of Dementia Detection: A Cluster Randomized Trial. Front Neurol. 2021 Jul 23;12:651826. doi: 10.3389/fneur.2021.651826. eCollection 2021. PMID 34367045